CLINICAL TRIAL: NCT03830320
Title: Preliminary Evaluation of [64Cu]FBP8 in Healthy Individuals and Subjects With Known or at Risk of Developing Thrombosis
Brief Title: Positron Emission Tomography (PET) Imaging of Thrombosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter Caravan, Professor of Radiology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P002385; R01HL109448 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-02-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; COVID-19; Cancer; Thrombosis
Keywords: PET-MRI
MeSH Terms: conditions — Atrial Fibrillation; COVID-19; Neoplasms; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (5):
- Healthy Volunteers (Active Comparator): Twenty (20) healthy adult subjects will be injected with [64Cu]FBP8 to establish the safety, whole body distribution, metabolism, pharmacokinetics, and radiation burden of the probe. All subjects will be imaged using PET/MR. Healthy subjects will undergo blood collection before, during, and after the scan. Healthy subjects will also undergo electrocardiogram before and after the scan. An interim review of the data will be conducted after the first six subjects receive the study agent and complete all safety assessments.
  Interventions: Drug: [64Cu]FBP8; Device: PET/MR; Procedure: Blood Collection; Procedure: Electrocardiogram
- Atrial Fibrillation Patients (Experimental): Thirty-five (35) patients with LAA thrombus documented by TEE will be injected with [64Cu]FBP8 and imaged for LAA thrombus with MR-PET. The TEE studies in these patients will be part of their routine clinical care. Thirty-five (35) patients with atrial fibrillation and negative TEE will be injected with [64Cu]FBP8 and imaged for LAA thrombus. Forty (40) patients with atrial fibrillation who are scheduled for TEE in the upcoming 14 days will be injected with [64Cu]FBP8 and imaged for LAA thrombus.
  Interventions: Drug: [64Cu]FBP8; Device: PET/MR
- COVID-19 Patients (Experimental): Thirty (30) COVID-19 patients will be injected with [64Cu]FBP8 and imaged for thrombi in the body.
  Interventions: Drug: [64Cu]FBP8; Device: PET/MR
- Cancer Patients (Experimental): Thirty (30) cancer patients will be injected with [64Cu]FBP8 and imaged for thrombi in the body.
  Interventions: Drug: [64Cu]FBP8; Device: PET/MR
- Other Thrombotic Condition Patients (Experimental): Fifty (50) patients with other thrombotic conditions will be injected with [64Cu]FBP8 and imaged for thrombi in the body.
  Interventions: Drug: [64Cu]FBP8; Device: PET/MR

INTERVENTIONS:
Drug: [64Cu]FBP8 — Injection of Copper-64 radiopeptide to detect thrombosis
  Other Names: 64Cu-FBP8
Device: PET/MR — Whole body imaging using Siemens mMR PET/MR scanner
  Other Names: PET-MR
Procedure: Blood Collection — A total of 9 cc of blood sampled before, during, and after imaging for clinical chemistry
  Arms: Healthy Volunteers
Procedure: Electrocardiogram — A standard 12-lead ECG will be obtained pre-and-post injection with radiotracer
  Other Names: ECG
  Arms: Healthy Volunteers

SUMMARY:
The purpose of the study is to evaluate a new radiotracer called 64Cu-FBP8 for PET-MR imaging of thrombosis. The tracer has the potential of detecting thrombosis anywhere in the body, for instance in the left atrial appendage of patients with atrial fibrillation, and thereby may provide a non-invasive alternative to the current standard-of-care methods.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. To evaluate the safety of [64Cu]FBP8 and its whole body distribution, metabolism, pharmacokinetics, and radiation burden in healthy volunteers.
2. To establish the accuracy of [64Cu]FBP8 -PET to detect left atrial thrombosis in patients with atrial fibrillation.
3. To explore the feasibility of [64Cu]FBP8 -PET to detect thrombosis in patients with COVID-19.
4. To explore the feasibility of [64Cu]FBP8 -PET to detect thrombosis in patients with cancer.
5. To explore the feasibility of [64Cu]FBP8 -PET to detect thrombosis in patients with known or suspicion of thrombus outside of the left atrial appendage.

ELIGIBILITY:
For Atrial Fibrillation Patient subjects:

* History of atrial fibrillation or paroxysmal atrial fibrillation;
* Retrospective enrollment: TEE to evaluate LAA within the last 14 days, provided the anticoagulation regimen the patient is on is not changed after the TEE. If a patient has a negative TEE and continues the same stable anti-coagulation regimen he/she is on, then it is extremely unlikely that a new thrombus will develop in the left atrial appendage within the next two weeks. Likewise, if a patient not taking any anti-coagulation has a thrombus in the left atrial appendage, then it is extremely unlikely that this thrombus will resolve spontaneously in the next 14 days if the patient continues not to take any anticoagulation. If the TEE leads to a change being made in the anticoagulation regimen (started/stopped/dose modified), then a time window of 72 hours from the TEE to PET imaging will be used. This scheme will ensure that the TEE can serve as an accurate gold standard;
* Prospective enrollment: TEE to evaluate LAA scheduled in upcoming 14 days;

For COVID-19 Patient subjects:

* Positive test for SARS-CoV-2 RNA detected by RT-PCR collected from the upper or lower respiratory tract analyzed by a certified lab with an FDA approved assay within the last month;
* Patient not requiring mechanical ventilation;

For Cancer Patient subjects:

• Patient is diagnosed with cancer;

For Other Patient subjects:

* Ultrasound- or CT-confirmed or high likelihood of thrombus (e.g., elevated D-dimer)
* Has not received thrombolytics

Exclusion criteria: A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Subjects less than 18 years of age;
* Electrical implants such as cardiac pacemaker or perfusion pump;
* Pregnant or breastfeeding (a negative STAT quantitative serum hCG pregnancy test is required for females having child-bearing potential before the subject can participate);
* Claustrophobic reactions;
* Subjects will be excluded if research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Unable to lie comfortably on a bed inside the PET scanner;
* Subjects under direct or indirect (i.e. same department as PIs) supervision of the principal investigator;
* Body weight over the weight limit for the moving table (> 300 lbs for the MRI table and >441 lbs for the CT table);
* Metallic or electric implants contraindicated for MR-PET scanning when applicable;
* Does not have the ability to give written informed consent.
* Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures);

Additional exclusion criteria for Atrial Fibrillation Patient subjects:

* Stroke within the last 3 months;
* Myocardial infarction within the last 3 months;
* Cardiac or major surgery within the last 3 months;
* History of chest pain within the last 6 weeks unless followed by a subsequent stress test or coronary angiography;
* History of syncope within the last 6 weeks;
* Heart rate persistently >120 bpm or persistently < 50 bpm;
* Presence of daytime pauses > 3s

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Complete blood count | 36 hours
  To model pharmacokinetics of [64Cu]FBP8 metabolism in healthy volunteers.
Target to Background Ratio LAA | 4 hours
  To determine the signal threshold of [64Cu]FBP8 that produces the highest accuracy of [64Cu]FBP8 -PET to detect left atrial thrombosis in patients with atrial fibrillation.
Target to Background Ratio | 4 hours
  To determine the signal threshold of [64Cu]FBP8 that produces the highest accuracy of [64Cu]FBP8 -PET to detect thrombosis in patients with known thrombus or suspicion of thrombus.
Time activity curve | 48 hours
  To evaluate human dosimetry and radiation burden in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Ciprian Catana, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Izquierdo-Garcia D, Desogere P, Philip AL, Mekkaoui C, Weiner RB, Catalano OA, Iris Chen YC, DeFaria Yeh D, Mansour M, Catana C, Caravan P, Sosnovik DE. Detection and Characterization of Thrombosis in Humans Using Fibrin-Targeted Positron Emission Tomography and Magnetic Resonance. JACC Cardiovasc Imaging. 2022 Mar;15(3):504-515. doi: 10.1016/j.jcmg.2021.08.009. Epub 2021 Oct 13. PMID 34656469